CLINICAL TRIAL: NCT02195973
Title: Phase IB Trial of LDE225 and Weekly Paclitaxel in Recurrent Platinum Resistant Ovarian Cancer
Brief Title: Phase IB Trial of LDE225 and Paclitaxel in Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Charles A Leath, III, MD, MSPH, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F140214007 (UAB 1357); 000505867 (Other: Office of Sponsored Programs)
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Ovarian Cancer
Keywords: ovarian cancer; platinum resistant; LED225; Sonidegib; Paclitaxel
MeSH Terms: conditions — Ovarian Neoplasms | interventions — sonidegib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Paclitaxel + LDE225 (Experimental): Patients will receive intravenous paclitaxel on days 1, 8, and 15 every 28 days (3 weeks on followed by one week off). This constitutes one cycle. in addition to the paclitaxel oral LDE225 will be taken daily. Dosages of each drug will vary according to the study cohort and phase. The study consists of six cycles of treatment followed by clinic visits every 2-3 months for up to two years.
  Interventions: Drug: LDE225

INTERVENTIONS:
Drug: LDE225 — After six cycles of weekly paclitaxel and LDE225, patients with a clinically beneficial response may be continued on weekly paclitaxel alone until disease progression.
  Other Names: Sonidegib (LDE225); Taxol (Paclitaxel)

SUMMARY:
The purpose of this study is to find out if a new drug, LDE225, is safe and has beneficial effects when combined with paclitaxel in women with platinum resistant ovarian cancer. Platinum resistant ovarian cancer refers to recurrent ovarian cancer that has undergone chemotherapy inclusive of a platinum compound (e.g. carboplatin or cisplatin).

DETAILED DESCRIPTION:
Ovarian cancer remains the deadliest gynecologic cancer with a fairly low long-term cure rate. LDE225 is a new type of drug that inhibits or blocks a pathway responsible for cancer cell growth. LDE225 is an investigational drug that has been used either solely or in combination with chemotherapy in other types of cancer but not in ovarian cancer. Research evidence suggests that by combining LDE225 and paclitaxel together, ovarian cancer cells may become more responsive to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent epithelial ovarian, fallopian tube or primary peritoneal carcinoma Histologic confirmation of the original primary tumor is required
* Papillary serous, endometrioid, clear cell, undifferentiated and mixed histologies
* Platinum resistant or refractory disease as per standard clinical and Gynecologic Oncology Group definition. Patients have had a treatment-free interval of less than 6 months from last platinum-based treatment to recurrence or progression during platinum based therapy
* Patients must have received at least one-prior platinum based chemotherapy regimen, to include cisplatin, carboplatin or other organoplatinum compound, for treatment of primary or recurrent ovarian, fallopian tube or primary peritoneal cancer
* Patients must have received a taxane as part of their prior treatment
* Measurable disease is required. By definition, measurable disease is at least one lesion that can be accurately measured in at least one dimension with the longest dimension to be recorded. Each lesion must be ≥ 20 mm when measured by conventional techniques, including palpation, plain x-ray, CT, MRI or ≥ 10 mm when measured by spiral CT imaging
* Patients must have one target lesion to be utilized in order to assess response per RECIST criteria
* ECOG Performance statuses of 0, 1, or 2
* Adequate organ function as evidenced by:

  1. Hematology: WBC ≥3.0 x 10^9/L; ANC ≥1.5 x 10^9/L; Platelets ≥100 x 10^9/L
  2. Renal function: Creatinine less than or equal to 1.5 x institutional upper limit of normal (ULN) or 24-hour clearance greater than or equal to 50 mL/min
  3. Hepatic function: Bilirubin ≤ 1.5 x ULN and ALT, SGOT and alkaline phosphatase ≤ 2.5 x ULN
  4. Plasma creatine phosphatase (CK) less than 1.5 x ULN
  5. Serum creatinine less than or equal to 1.5 x ULN or 24-hour clearance greater than or equal to 50 mL/min
* Signed informed consent.
* Female patients of any ethnic group. Female patients must be surgically sterile, postmenopausal (no menses for at least one year), or using medically approved method of contraception (excluding rhythm, withdraw or abstinence)
* Age greater than or equal to 19
* Recovery from effects of any recent surgery, chemotherapy and/or radiation

  1. No evidence of active infection requiring antibiotic therapy
  2. Hormonal therapy being utilized, as an anti-neoplastic treatment must be discontinued at least one week prior to study entry. Hormonal replacement therapy for symptom management is allowed
  3. Any prior therapy directed at the malignancy including biologic or immunologic agents, must have be discontinued at least three weeks prior to study entry

Exclusion Criteria:

* Patients with pathology demonstrating mucinous, carcinosarcoma or low malignant potential tumor histology are excluded. In addition, non-ovarian malignancies, malignant germ cell or stromal tumors are also excluded
* Previous or concurrent malignancies at other sites within the last 5 years, with the exception of in situ carcinoma of the cervix and adequately treated basal cell carcinoma or squamous cell carcinoma of the skin. In addition, patients with prior or concomitant, based on hysterectomy, Stage IA endometrial adenocarcinoma with less than 3 mm depth on invasion, absence of lymphovascular space invasion and absence of grade 3, papillary serous or clear cell histology are allowed
* Patients with prior radiation to the abdominal cavity or pelvis are excluded
* Patients unable to take oral drugs or with lack of physical integrity of the upper gastrointestinal tract or known malabsorption syndromes
* Patients who have previously been treated with systemic sonidegib (LDE225) or with other Hh pathway inhibitors
* Serious concomitant illness including but not limited to: uncontrolled diabetes mellitus, dementia, active infection (including HIV infection) requiring IV or oral antibiotics and psychiatric illness and/or other uncontrolled medical conditions which may preclude compliance with study protocol
* Patients who have neuromuscular disorder (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis and spinal muscular atrophy) or are on concomitant treatment with drugs that are recognized to cause rhabdomyolysis, such as HMG CoA inhibitors (statins), clofibrate and gemfibrozil, and the cannot be discontinued at least 2 weeks prior to starting sonidegib treatment. If it is essential that the patient remain on a statin to control hyperlididemia, only pravastatin may be used with extra caution
* Patients who are planning on embarking on a new strenuous exercise regimen after initiation of study treatment. Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided whilst on sonidegib treatment
* Patients who have taken part in an experimental drug study within 4 weeks or 5 half-lives, whichever is longer, of initiating treatment with sonidegib
* Patients who are receiving other anti-neoplastic therapy (e.g. chemotherapy, targeted therapy or radiotherapy) concurrently or within 2 weeks of starting treatment with sonidegib
* Peripheral Neuropathy of NCI-CTC (National Cancer Institute-Common Toxicity Criteria) grade greater than or equal to 2
* Impaired cardiac function or clinically significant heart disease, including any one of the following:

  1. Angina pectoris within 3 months
  2. Acute myocardial infarction within 3 months
  3. QTcF > 470 msec on the screening ECG
  4. A past medical history of clinically significant ECG abnormalities or a family history of prolonged QT-interval syndromes
  5. Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>5 mIU/mL)
* Patients who are not willing to apply highly effective contraception during the study and through the duration as defined below after the final dose of study treatment

  a. Women of childbearing potential defined as all women physiologically capable of becoming pregnant. Must use highly effective contraception during the study and through 20 months after the final dose of study treatment. Highly effective contraception is defined as either:
  1. Total abstinence: When this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  2. Sterilization: Patient has had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman had been confirmed by follow- up hormone level assessment
  3. Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female study patients, the vasectomized male partner should be the sole partner for that patient
  4. Use a combination of the following (both a + b):

     1. Placement of a non-hormonal intrauterine device (IUD) or non- hormonal intrauterine system (IUS)
     2. Barrier method of contraception: Condom or occlusive cap (diaphragm or cervical vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

        Note: Hormonal contraception methods (e.g. oral, injected, implanted) are not allowed as it cannot be ruled out that the study drug decreases the effectiveness of hormonal contraception.

        Note: Women are considered post-menopausal and not child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels >40 mIU/mL and estradiol <20 pg/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six week ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* History of hypersensitivity to paclitaxel
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Patients who are receiving treatment with medications known to be moderate and strong inhibitors or inducers of CYP3A4/5 or drugs metabolized by CYP2B6 or CYP2C9 that have narrow therapeutic index, and that cannot be discontinued before starting treatment with sonidegib. Medications that are strong CYP3A4/5 inhibitors should be discontinued at least 7 days and strong CYP3A/5 inducers for at least 2 weeks prior to starting treatment with sonidegib

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-12-10 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Safety of weekly paclitaxel + LDE225 treatment | up to 2 years
  Safety of weekly paclitaxel and LDE225 treatment in patients with recurrent, platinum-resistant ovarian adenocarcinoma will be monitored by physical exams, review of adverse events, and laboratory studies.
Assessment of toxicities | up to 2 years
  Assessment of toxicity will be performed using the National Cancer Institute Common Toxicity Criteria version 4.03.

SECONDARY OUTCOMES:
Optimal dose of LDE225 with paclitaxel | 6 months
  The maximum tolerated dose and dose-limiting toxicities of weekly paclitaxel and daily LDE225 will be determined from laboratory tests on blood collected one to two times each cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Leath, III, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No